CLINICAL TRIAL: NCT02354053
Title: A Phase IV, Multicentre Randomized Prospective Open Label Study to Evaluate Whether Switching From Current cART to Triumeq in Addition to Adherence Support Will Enhance Virologic Control and Adherence in Vulnerable Populations Relative to Adherence Support Alone
Brief Title: Evaluation of Switching From Current cART to Triumeq With Adherence Support Will Enhance HIV Control in Vulnerable Populations
Acronym: TRIIADD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: ViiV Healthcare (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Marina Klein, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTN286
Record Dates: First submitted 2015-01-27; First posted 2015-02-03 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: HIV Infections
Keywords: HIV; Triumeq; vulnerable populations
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Current ART (Active Comparator): Current ART + adherence support
  Interventions: Behavioral: Adherence support + current ART
- Triumeq (Experimental): Triumeq + adherence support
  Interventions: Drug: Switch to Triumeq; Behavioral: Adherence support + current ART

INTERVENTIONS:
Drug: Switch to Triumeq
  Arms: Triumeq
Behavioral: Adherence support + current ART

SUMMARY:
Modern antiretroviral therapeutic regimens offer a vast array of choice that permits tailored therapy for HIV patients. While modern regimens have improved the rates of virologic suppression overall and reduced adverse effects of antiretroviral treatment, an important sub-group of HIV infected persons is unable to maintain adherence to their treatment regimens, fail to achieve long term virologic control and remain at risk for HIV related disease progression and transmission of HIV infection.

Hypothesis: switching from current cART regimen to a Triumeq based regimen combined with adherence support will improve the rate of HIV suppression in vulnerable populations non-adherent to the their current cART as determined by the achievement of HIV-1 RNA < 50 copies/mL at Week 24 post randomization.

DETAILED DESCRIPTION:
Primary objectives:

To determine if switching from current cART regimen to a Triumeq based regimen combined with adherence support will improve the rate of HIV suppression in vulnerable populations non-adherent to the their current cART as determined by the achievement of HIV-1 RNA < 50 copies/mL at Week 24 post randomization.

Secondary objectives:

In vulnerable populations non-adherent to their current cART:

(i) To determine if switching from current cART to a Triumeq based regimen will improve the average adherence of patients compared to maintaining current cART, measured at 24 weeks post randomization.

(ii) To determine if adherence is maintained over the long term (up to 72 weeks) in subjects receiving Triumeq (iii) To evaluate the effect of switching to Triumeq on control of HIV infection (as measured by HIV viral load and CD4 cell counts) up to 72 weeks (iv) To determine the safety of using Triumeq with respect to risk for the emergence of HIV drug resistance.

(vi) To assess the safety and tolerability (including hepatic function and metabolic profiles) of switching from current cART regimen to Triumeq up to 72 weeks.

(vi) To evaluate if switching to Triumeq will be cost effective from a societal prospective

Study Population:

We will recruit from 14 CTN-affiliated sites across Canada.

All patients recruited into the trial will be adults aged over 18 years old with documented HIV infection (ELISA with western blot confirmation) and with negative HLA-B5701 testing. Prescribed ART may include any DHHS recommended or alternative regimens, which the treating physician considers, is appropriate for their patient (except dolutegravir) for at least 6 months. Subjects will have evidence of non-adherence to current ART regimen defined as:

* HIV RNA ≥400 copies/ml at least once in last 12 months
* Absence of evidence of resistance to any component of the current regimen or Triumeq
* Viremia not explained by normal viral decay after initiating ART We anticipate that many of recruited subjects will comprise people who inject drugs, Aborginal persons and persons from ethnocultural communities however recruitment will not be limited to these groups as others may be enrolled provided they meet the inclusion criteria.

Study design:

A randomized, prospective, open-label study. Patients will be randomized 1:1 to switch to Triumeq vs. to remain on current cART. Both groups will receive adherence support. Those randomized to maintain current cART will be permitted to switch to Triumeq after 24 weeks.

Sample size:

N = 100 100 patients (50/arm) will provide 80% power to detect a 25% difference in virologic suppression rates between the two arms at 24 weeks. While this difference is large, for the population we are targeting we consider that an improvement in virologic suppression rates of at least this amount would be required to be clinically meaningful.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults greater than or equal to 18 years of age.
2. Prescribed cART that may include any DHHS recommended or alternative regimens, which the treating physician considers, is appropriate for their patient with the exception of dolutegravir
3. Evidence of non-adherence to current ART regimen defined as:

   1. HIV RNA ≥400 copies/ml at least once in last 12 months
   2. Absence of resistance to current regimen
   3. Viremia not explained by normal viral decay after initiating ART
4. Documentation that the subject is negative for HLA-B*5701 allele
5. Signed informed consent prior to screening.
6. Women who are suspected, planning to become or pregnant or breastfeeding must have a negative pregnancy test at screening and Day 1 and agree to use the following approved methods of birth control while on study.

   A female, may be eligible to enter and participate in the study if she:
   1. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
   2. is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:

      * Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all study medications;
      * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
      * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion
      * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
      * Approved hormonal contraception
      * Any other method with published data showing that the expected failure rate is <1% per year.

   Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of Triumeq.
7. Heterosexual men should use at least one barrier method of contraception (e.g. condom)

Exclusion Criteria:

1. Not meeting inclusion criteria
2. Women who are pregnant or breastfeeding
3. Any evidence of an active Centers for Disease and Prevention Control (CDC) Category C disease25 except cutaneous Kaposi's sarcoma not requiring systemic therapy
4. Subjects with moderate to severe hepatic impairment (Class B or C) as determined by Child-Pugh classification
5. Anticipated need for Hepatitis C virus (HCV) therapy during the study
6. Chronic hepatitis B infection (defined as HBsAg positive)
7. History or presence of allergy or intolerance to the study drugs or their components or drugs of their class
8. Any evidence of viral resistance to 3TC, abacavir or integrase inhibitors or to any component of the current regimen based on the presence of primary resistance-associated mutations for these drugs26 on any available historical resistance test.
9. Any evidence of viral resistance to 3TC, abacavir or integrase inhibitors or to any component of the current regimen based on the presence of primary resistance-associated mutations for these drugs26 on a screening genotype for patients with HIV RNA ≥400 copies/ml .
10. Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study
11. Alanine aminotransferase (ALT) greater than 5 times the upper limit of normal, OR ALT greater than or equal to3 times the upper limit of normal and bilirubin greater than or equal to1.5 times the upper limit of normal (with greater than 35% direct bilirubin)
12. Creatinine clearance of less than 50 mL/min via Cockroft-Gault method
13. Concomitant medications, dofetilide and immunosuppressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-11; Primary Completion 2018-07-03 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of the Switch from ART to Triumeq with adherence support as determined by the achievement of HIV-1 RNA < 50 copies/mL at Week 24 post randomization. | 24 weeks
  To determine if switching from current cART regimen to a Triumeq based regimen combined with adherence support will improve the rate of HIV suppression in vulnerable populations non-adherent to the their current cART.

SECONDARY OUTCOMES:
Improve of average adherence | 24 weeks
  To determine if switching from current cART to a Triumeq based regimen will improve the average adherence of patients compared to maintaining current cART, measured at 24 weeks post randomization. We will use a set of questionnaires:
  * HIV treatment knowledge questionnaire: this questionnaire will help to identify any patients that may need psycho-education regarding HIV treatment (patients who failed to answer to any knowledge item)
  * Experience of Close Relationships (ECR-short)
  * Patient Health Questionnaire (PHQ9).
  * Alcohol: Audit C:
  * Drug abuse Drug Use Disorders Identification Test (DUDIT)27.
  * Quality of life using the EuroQoL EQ-5D tool
  * HIV Cost and Services Utilization Study questionnaire.
Maintaining Adherence over the time | 72 weeks
  To determine if adherence is maintained over the long term (up to 72 weeks) in subjects receiving Triumeq

CONTACTS AND LOCATIONS:
Overall Officials: Marina Klein, MD, Principal Investigator — Chronic Viral Illness Service
Locations (1):
- Chronic Viral Illness Service, Montreal, Quebec, Canada